CLINICAL TRIAL: NCT04981847
Title: Ensuring the Cultural Relevance of Dietary Guidelines Diet Patterns Among African Americans: Increasing Dietary Quality and Reducing Type 2 Diabetes Risk
Brief Title: The Dietary Guidelines 3 Diets Study
Acronym: DG3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00105836
Record Dates: First submitted 2021-07-27; First posted 2021-07-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to participant group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- US Healthy Diet (Experimental): Participants in this group will be assigned to follow the Healthy US dietary pattern as presented by the US Dietary Guidelines. As described here https://www.nia.nih.gov/health/usda-food-patterns: This eating pattern is based on the types and amounts of foods Americans typically consume. The main types of food in this eating pattern include a variety of vegetables; fruits; whole grains; fat-free or low-fat dairy; seafood, poultry, meat, and eggs; and nuts, seeds, and soy products.
  Interventions: Behavioral: Dietary Intervention Meetings
- Mediterranean diet (Experimental): Participants in this group will be assigned to follow the Mediterranean dietary pattern as presented by the US Dietary Guidelines. As described here https://www.nia.nih.gov/health/usda-food-patterns: This eating pattern contains more fruits and seafood and less dairy than the Healthy U.S.-Style Eating Pattern. There is also less calcium and vitamin D because it includes fewer dairy foods.
  Interventions: Behavioral: Dietary Intervention Meetings
- Vegetarian diet (Experimental): Participants in this group will be assigned to follow the Vegetarian dietary pattern as presented by the US Dietary Guidelines. As described here https://www.nia.nih.gov/health/usda-food-patterns: This eating pattern contains no meat, poultry, or seafood. Compared with the Healthy U.S.-Style Eating Pattern, it contains more soy products, eggs, beans and peas, nuts and seeds, and whole grains.
  Interventions: Behavioral: Dietary Intervention Meetings

INTERVENTIONS:
Behavioral: Dietary Intervention Meetings — Participants will attend classes once per week for 3 months.

SUMMARY:
The goal of this project is to use a two-stepped study to examine both the adoption of the three dietary patterns as presented by the United States Dietary Guidelines (USDG) and testing of a refined, culturally tailored one-year intervention examining the three diet patterns. For this study, African American adult participants with overweight/obesity and ≥three type 2 diabetes (T2DM) risk factors will be recruited to participate in this two-step study. This present study is for our Step 1: formative pilot work to culturally-tailor a dietary intervention of the three healthy eating patterns presented by the USDG for 12 weeks: 1) U.S.-Style, 2) Mediterranean, or 3) Vegetarian.

DETAILED DESCRIPTION:
The U.S. Dietary Guidelines (USDG) form the basis of federal nutrition programs and policy and provide valuable guidance to health initiatives and industries. The updated 2015 USDG moved away from a focus on individual nutrients to a greater focus on dietary patterns. The USDG state that healthy eating goals can be met through a variety of dietary patterns, but present healthy diet in three main ways: 1) Healthy U.S.-Style Eating Pattern, 2) Healthy Mediterranean-Style Eating Pattern, and 3) Healthy Vegetarian Eating Pattern. Currently, US adults are falling short of the nutrition recommendations (fruit/vegetable intake, greens/beans, whole grains, etc.) set forth by the USDG and measured by the Healthy Eating Index (HEI). While the USDG are the basis of nutrition guidelines, the research informing these dietary pattern recommendations has largely been drawn from observational studies among mostly white populations. In addition, there has been very limited cultural tailoring of these dietary patterns that would ensure that these diets are acceptable to diverse populations, in particular, African Americans (AAs) living in the south, who experience a disproportionate burden of chronic disease, especially type 2 diabetes (T2DM). Currently, US adults are not meeting nutrition recommendations (fruit/vegetable, whole grains, etc.) set forth by the USDG and measured by the Healthy Eating Index (HEI).

For the present study, AA adult participants with overweight/obesity and ≥three T2DM risk factors will be recruited to participate in the following aims:

Aim 1: Conduct a 3-month randomized trial among AAs comparing adoption of the 3 dietary patterns [1) US, 2) Med, or 3) Veg] using existing materials from the USDG and examine differences in diet quality (HEI) and T2DM risk factors (weight, HgbA1c).

Aim 2: Drawing on participants' experiences in Aim 1, conduct qualitative work to refine and culturally tailor the dietary pattern intervention for an AA audience.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* BMI between 25- 49.9 kg/m2
* self-identify as African American
* live in the Columbia, SC area
* be able to attend all monitoring visits
* be willing to be randomized to either condition and be re-randomized if non-responsive
* be free of major health or psychiatric diseases, drug or alcohol dependency, thyroid conditions, diabetes, or pregnancy

Exclusion Criteria:

* should not be pregnant (or have been pregnant in the last 6 months), anticipating on becoming pregnant in the next 24 months, or currently breastfeeding

  o Women who are pregnant should not be pursuing weight loss and should be under the direct care of a physician. Therefore women who are pregnant or who are anticipating they might be pregnant should not participate in this study. If a woman becomes pregnant during the study, she will be advised to consult with her healthcare provider and will be dropped from the weight loss study.
* should be free of an eating disorder as screened by the Eating disorder Screen for Primary care [ESP]. (If a participant has an eating disorder, they will be given contact information for the eating disorder clinic at the University of South Carolina)
* no current participation in a weight loss program or taking weight loss medications (although participants may be trying to lose weight on their own)
* no recent or planned bariatric surgery
* no recent weight loss (>10 lbs in the last 6 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Dietary quality | 3 months
  Dietary quality as assessed by the Healthy Eating Index
Body weight | 3 months
  Changes in body weight
Hemoglobin A1c | 3 months
  Changes in HgbA1c over 3 months

SECONDARY OUTCOMES:
Blood pressure | 3 months
  changes in systolic and diastolic blood pressure over 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

REFERENCES:
- [Derived] Turner-McGrievy G, Wirth MD, Okpara N, Jones M, Kim Y, Wilcox S, Friedman DB, Sarzynski MA, Liese AD. Similar changes in diet quality indices, but not nutrients, among African American participants randomized to follow one of the three dietary patterns of the US Dietary Guidelines: A secondary analysis. Nutr Res. 2024 Nov;131:27-38. doi: 10.1016/j.nutres.2024.09.005. Epub 2024 Sep 7. PMID 39366028
- [Derived] Turner-McGrievy GM, Wilson MJ, Carswell J, Okpara N, Aydin H, Bailey S, Davey M, Hutto B, Wilcox S, Friedman DB, Sarzynski MA, Liese AD. A 12-Week Randomized Intervention Comparing the Healthy US, Mediterranean, and Vegetarian Dietary Patterns of the US Dietary Guidelines for Changes in Body Weight, Hemoglobin A1c, Blood Pressure, and Dietary Quality among African American Adults. J Nutr. 2023 Feb;153(2):579-587. doi: 10.1016/j.tjnut.2022.11.020. Epub 2022 Dec 23. PMID 36894249